CLINICAL TRIAL: NCT03785197
Title: Effects of a Clinical Dietary Intervention During Inpatient Treatment (Modified Fasting in Metabolic Syndrome, Osteoarthritis of the Hip or Knee, Rheumatoid Arthritis and Fibromyalgia)
Brief Title: Effects of a Clinical Dietary Intervention During Inpatient Treatment
Acronym: FASTA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: FASTA
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Metabolic Syndrome; Osteoarthritis, Hip; Osteoarthritis, Knee; Rheumatoid Arthritis; Fibromyalgia
Keywords: fasting; natural therapies; prolonged fasting
MeSH Terms: conditions — Metabolic Syndrome; Osteoarthritis, Hip; Osteoarthritis, Knee; Arthritis, Rheumatoid; Fibromyalgia; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prolonged modified fasting — The prolonged modified fasting is a dietary intervention with abstinence from solid foods and a caloric intake of 100-400 kcal through juices and vegetable broths

SUMMARY:
The purpose of the study is a scientific and prospective documentation of the clinical effects of an inpatient treatment at the Immanuel Hospital of Berlin, in the department for complementary and integrative medicine, with the use of a modified fasting regime. A pre- and post- as well as group comparisons are planned. Patients that are admitted to the inpatient department for metabolic syndrome, osteoarthritis of the hip or knee, rheumatoid arthritis and fibromyalgia will be enrolled in the study.

DETAILED DESCRIPTION:
At the beginning, during and at the end of the treatment at the inpatient department routine blood parameters, anthropometric parameters and certain scores and parameters specific to the different conditions will be measured. Questionnaires will be filled out by patients before and after the treatment as well as 3, 6 and 12 months after leaving the inpatient department.

ELIGIBILITY:
Inclusion Criteria:

* The patient is consents to participating in the trial during the first 24h of his or her stay in the inpatient naturopathic department of the Immanuel Hospital.
* Written informed consent is given
* The referral diagnosis is one of the following: diabetes mellitus type 2/metabolic syndrome, osteoarthritis of the hip, osteoarthritis of the knee, rheumatoid arthritis, fibromyalgia.

Exclusion Criteria:

* Language barries to understanding the instructions of the study personnel
* Dementia or other strong cognitive impairment
* Pregnant or lactating women
* Taking part in another study at the same time

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regular hospitalised patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; The FIQ is scored in such a way that a higher score indicates a greater impact of the syndrome on the person. Each of the 10 items has a maximum possible score of 10. Thus the maximum possible score is 100. The average FM patient scores about 50, severely afflicted patients are usually 70 plus.
Disease Activity Score 28 (DAS 28) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire with Clinical Examination; Change from Baseline in the DAS-28, range from 2.0 to 10.0 while higher values meaning a higher disease activity and below of 2.6 meaning remission
Health Assessment Questionnaire (HAQ) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; Change from Baseline in the HAQ, range from 0 to 3 while higher values meaning a higher grade of disability
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire consisting of 24 items divided into 3 subscales: Pain (5items), Stiffness (2 items), Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher values meaning a higher grade of disability.
Summary of Diabetes Self Care Activities Measure (SDSCA) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; 11 items with each item scored on a scale of 0-7.

SECONDARY OUTCOMES:
Pain on Visual Analogue Scale (VAS) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire
Hospital Anxiety and Depression Scale (HADS) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; HADS: Assessing full scale, range 0-42, lower score meaning a better outcome
Perceived Stress Scale (PSS) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; Change from Baseline in the PSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items while higher values meaning a higher grade of perceived stress.
Quality of Life (WHO-5) | Change Baseline, 2 weeks, 3 months, 6 months, 12 months
  Questionnaire; Change from Baseline in the WHO-5, range from 0 to 100 % while higher values meaning a higher grade of well-being
Body-Mass-Index (BMI) | Change Baseline, 2 weeks
  Anthropometry
Blood pressure | Change Baseline, 2 weeks
  Measuring systolic and diastolic blood pressure in mmHg
24h-Blood pressure | Change Baseline, 2 weeks
  Measuring systolic and diastolic blood pressure with Device "Mobil-O-Graph"
Blood count | Change Baseline, 2 weeks
  Laboratory test
Glomerular filtration rate (GFR) | Change Baseline, 2 weeks
  Laboratory test
Blood lipids | Change Baseline, 2 weeks
  triglycerides (mmol/L), total cholesterol (mmol/L), LDL (mmol/L), HDL (mmol/L), fasting glucose (mmol/L)
CRP | Change Baseline, 2 weeks
  CRP in milligram per liter (mg/L)
Liver enzymes (GOT, GPT) | Change Baseline, 2 weeks
  Hepatic transaminases (GPT, GOT in U/L)
Stepcounter | Change Baseline, 2 weeks
  With Device "Everion"
Heart Rate Variability | Change Baseline, 2 weeks
  With Device "Faros 180"
Heart Rate | Change Baseline, 2 weeks
  With Device "Everion"
Blood Oxygenation | Change Baseline, 2 weeks
  With Device "Everion"

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Study Principal Investigator
Locations (1):
- Immanuel Hospital, Wannsee, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koppold DA, Kandil FI, Muller A, Guttler O, Steckhan N, Meiss S, Breinlinger C, Nelle E, Rajput Khokhar A, Jeitler M, Hanslian E, Fischer JM, Michalsen A, Kessler CS. Effects of Prolonged Medical Fasting during an Inpatient, Multimodal, Nature-Based Treatment on Pain, Physical Function, and Psychometric Parameters in Patients with Fibromyalgia: An Observational Study. Nutrients. 2024 Apr 4;16(7):1059. doi: 10.3390/nu16071059. PMID 38613092